CLINICAL TRIAL: NCT06678399
Title: Phase 1B/2 Clinical Trial Assessing the Safety, Tolerability and Preliminary Efficacy of the Allogeneic Placental Mesenchymal Cells for the Preemptive Treatment of Patients At Risk for Acute Kidney Injury Following Cardiac Surgery
Brief Title: Phase 1B/2 Clinical Trial Assessing the Safety, Tolerability and Preliminary Efficacy of the Intravenous Administration of Allogeneic Placental Mesenchymal Cells for the Preemptive Treatment of Patients At Risk for Acute Kidney Injury Following Cardiac Surgery
Acronym: MesAKI
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kelifarma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KELI-101
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Preemptive Therapy of Patients At Risk for Acute Kidney Injury Following Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Low dose (Experimental)
  Interventions: Drug: KELI-101
- High dose (Experimental)
  Interventions: Drug: KELI-101
- Historical matched-control group (No Intervention)
- Best dose (Experimental)
  Interventions: Drug: KELI-101
- Placebo (Placebo Comparator)
  Interventions: Other: Vehicle (placebo)

INTERVENTIONS:
Drug: KELI-101 — KELI-101 consists of ex vivo expanded placental mesenchymal stromal cells (PMSCs) in a 10% cryopreservation solution.
  Arms: Best dose; High dose; Low dose
Other: Vehicle (placebo) — Plasmalyte
  Arms: Placebo

SUMMARY:
This clinical trial is designed to evaluate KELI-101 versus placebo for the prevention of acute kidney disease leading to chronic kidney disease in subjects at high risk for acute kidney injury following cardiac surgery. Half of the participants will receive KELI-101, while the other half will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

Pre-operative

1. Age ≥ 45 years at screening.
2. Weigh at least 50 kg and maximum 150 kg to participate in the study and must have a body mass index (BMI) below 40; BMI = Body weight (kg) / [Height (m)]2.
3. Estimated kidney volume within normal ranges (110-190 ml for male and 90-150 ml for female, ultrasound method, ellipsoid formula)
4. High risk for AKI post CABG development as assessed by investigator e.g., >9 points by Acute Renal Failure after Cardiac Surgery (Thakar Score, Cleveland Clinic Score)
5. At screening, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position. Sitting vital signs should be within the following ranges:

   1. oral body temperature between 35.0-37.5 °C
   2. blood pressure (systolic 100-160 mmHg, diastolic < 100 mmHg)
   3. pulse rate (50-100/min) stable with or without medication(s) as per Investigator assessment.
6. Have a pre-operative (baseline) SCr and uNGAL collected within 30 days of surgery (if multiple laboratory results are available within this time window, the most recent SCr and uNGAL values before surgery will be used to establish the baseline)
7. No known change (increase or decrease) in SCr of ≥25% and uNGAL >200% at screening visit compared to a previous value not older than 6 weeks as documented by a local laboratory using standard assay methodology.
8. Willing and able to comply with visit schedule and study procedures including post-hospitalization discharge follow-up.
9. Ability to give informed consent or have a legally acceptable representative do so for them.

   Peri-operative
10. Non-emergent cardiovascular surgery utilizing CPB with >1 hr duration time. Post-operative
11. ≥ 200% rise in uNGAL and uNGAL/Cr from baseline AND above cut-off of 34 ng/mg Cr (in nonCKD patients) within 4 hours of removal from CPB [the timeline and cut-off values TBD after Phase 1 (IA1)]

Exclusion Criteria:

Pre-operative

1. eGFR at screening <30 mL/min/1.73 m2 (calculated using CKD-EPI 2021 equation), or on dialysis.
2. Currently receiving renal replacement therapy.
3. Patients with bleeding risk at screening. The Investigator should make this determination in consideration of the participant's medical history and/or clinical or laboratory evidence of any of the following:

   1. History of bleeding with suspected or confirmed bleeding disorder or any other high risk for bleeding in the opinion of the investigator.
   2. Thrombocytopenia: platelet count< 100x109/L
   3. Platelet dysfunction: e.g., ADP-induced platelet aggregation lower than 60 %.
   4. Pre-existing coagulation factor deficiency: including, but not limited to, fibrinogen < 2.5-2.8 g/L
4. Any emergency surgeries performed less than 30 days before screening, including aortic dissection and/or significant congenital heart defects.
5. Class IV heart failure according to the functional classification of the New York Heart Association (NYHA).
6. Left ventricular ejection fraction < 30% (based on the last available cardiac ultrasound).
7. Scheduled to undergo cardiac surgery off CPB or with hypothermic circulatory arrest.
8. Cardiogenic shock or hemodynamic instability within four weeks before surgery, requiring inotropes or vasopressors or mechanical devices such as intra-aortic balloon counter-pulsation (IABP).
9. Have received cardiopulmonary resuscitation (CPR) within 30 days before cardiac surgery.
10. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or until the expected pharmacodynamic (PD) effect has returned to baseline, whichever is longer; or longer if required by local regulations.
11. Patients who are post-nephrectomy
12. Uncontrolled diabetes (glycolyzed HGB <7 or another cut-off as per clinical guidelines for a particular patient)
13. Have ongoing sepsis, history of sepsis or uncontrolled infection within the past 8 weeks or untreated diagnosed infection before screening visit. Sepsis is defined as the presence of a confirmed pathogen, along with fever or hypothermia and hypoperfusion or hypotension.
14. Prescribed nephrotoxic medicines (aminoglycosides, glycopeptides, radiocontrast or other agents) within the past week, leading to increased sCr >25%
15. Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
16. Pregnant or nursing (lactating) women
17. Women of child-bearing potential are defined as all women physiologically capable of becoming pregnant unless they are using highly effective methods of contraception while taking study treatment and until the end of the study. Highly effective contraception methods include:

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Female bilateral tubal ligation, female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or total hysterectomy at least six weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
    3. Male sterilization (at least 6 months before screening). For female participants in the study, the vasectomized male partner should be the sole partner for that participant.
    4. Use of oral (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example, hormone vaginal ring or transdermal hormone contraception Peri-, postoperative
18. Anemia and hemotransfusion.
19. History of oncological disorders.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAE) | From KELI -101 administration up to Day 90
  To assess the acute and middle-term toxicity of the intrarenal arterial administration of KELI -101
Ratio of the acute kidney disease (AKD) leading to chronic kidney disease (CKD) | From baseline to Day 90
  To assess the effect of KELI -101 on AKD leading to CKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo

SECONDARY OUTCOMES:
Adverse events (AE) and adverse drug reactions (ADRs) | From KELI -101 administration up to Day 90
  To assess tolerability and all AE (related or not related to study drug) after IRA administration of KELI -101
Serious AE (SAE) and Serious ADRs (SADRs) | From KELI -101 administration up to Day 90
  To assess all serious AE (related or not related to study drug) after IRA administration of KELI -101
Ratio of the highest SCr value within 6 days post-dose versus baseline | From baseline to Day 7
  To assess the effect of KELI -101 on SCr level, versus mean matched historical control SCr level
AKI stages 1, 2 and 3 as defined by modified AKI Network criteria | From baseline to Day 7
  To assess the effect of KELI -101 on the incidence and severity of AKI in high-risk patients undergoing major cardio-vascular surgery, versus mean matched historical control SCr level
  For historical control:
  To assess the incidence and severity of AKI in high-risk patients undergoing major cardiovascular surgery in relation to preoperative Scr levels.
Ratio of the duration of AKI/AKD at Day 28 | From baseline to Day 28
  To assess the effect of KELI -101 on duration of AKI/AKD
Ratio of incidence and duration of renal replacement therapy (RRT) Day 28 | From baseline to Day 28
  To assess the effect of KELI -101 on incidence and duration of RRT
Occurrence of major adverse kidney event (MAKE) at Day 7/10/30/90 (MAKE7/10/30/90) | From Day 7 to Day 90
  To assess the effect of KELI -101 on Major Adverse Kidney Events composite (MAKE7/10/30/90)
Occurrence of major adverse reno cardiovascular event at Day 7/10/30/90 (MARCE7/10/30/90) | From Day 7 to Day 90
  To assess the effect of KELI -101 on Major Adverse Reno Cardiovascular Events composite (MARCE7/10/30/90)
Ratio of the AKI leading to CKD | From baseline to Day 90
  To assess the effect of KELI -101 on incidence of AKI to CKD transition;
Ratio of duration of stay in ICU | From baseline to discharge from ICU
  To assess the effect of KELI -101 on length of ICU-stay
Ratio of incidence and completeness of recovery of AKI/AKD at Day 90 | From baseline to Day 90
  To assess the effect of KELI -101 on complete or partial recovery and non-recovery of AKI/AKD
Ratio of CKD severity as per eGFR and albuminuria at Day 90 | Day 90
  To assess the effect of KELI -101 on sustained decline in renal function
For matched control cohort: Increased uNGAL and uNGAL/Cr in patients that develop AKI | Timepoints of 3 Pre-CPB (D-30, D-10 to D-3 and D-1) and 5 (6) after CPB initiation: (CPB-H2, CPB-H3-4, CPB-H5-6, CPB-H9-12, (CPB-H24), and one immediately post-CPB time point (+5 to 15 min), optional
  To assess the magnitude of Increased uNGAL and uNGAL/Cr values in urine in patients that develop AKI as compared to those without developed AKI (21 patients for AKI patients and 10 non-AKI patients' cohorts)
For matched control cohort: Prognostic value of increased uNGAL and uNGAL/Cr, duration, and area under curve in patients that develop AKI as compared to patients that do not develop AKI | Timepoints of 3 Pre-CPB (D-30, D-10 to D-3 and D-1) and 5 (6) after CPB initiation: (CPB-H2, CPB-H3-4, CPB-H5-6, CPB-H9-12, (CPB-H24), and one immediately post-CPB time point (+5 to 15 min), optional
  To assess the magnitude of Increased uNGAL and uNGAL/Cr values, duration, and area under curve in patients that develop AKI as compared to those without developed AKI (21 patients for AKI patients and 10 non-AKI patients' cohorts)
Ratio of the acute kidney disease (AKD) at Day 10 leading to chronic kidney disease (CKD) at Day 90 | From baseline to Day 90
  To assess the effect of KELI -101 on AKD leading to CKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo
Ratio of incidence and duration of RRT Day 28 | From baseline to Day 28
  To assess the effect of KELI -101 on incidence and duration of RRT
Occurrence of major adverse kidney event at Day 90 (MAKE90) | Day 90
  To assess the effect of KELI -101 on the incidence of AKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo
Occurrence of major adverse kidney event at Day 30 (MAKE30) | Day 28+2 (Phone call)
  To assess the effect of KELI -101 on the incidence of AKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo
Occurrence of individual components of the MAKE criteria at Days 30 or 90 | Day 28+2 (Phone call)
  To assess the effect of KELI -101 on the incidence of AKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo
Occurrence of individual components of the MARCE criteria at Days 7/10/30/90 | From Day 7 to Day 90
  To assess the effect of KELI -101 on the incidence of AKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo
CKD severity as per eGFR and albuminuria at Day 90 | Day 90
  To assess the effect of KELI -101 on sustained decline in renal function